CLINICAL TRIAL: NCT06552715
Title: Pilot Clinical Study on the Efficacy of a Flexible Hydroxyapatite-Based Composite for the Regeneration of Jaw Bone Defects
Brief Title: Pilot Study on the Effectiveness of a Flexible Hydroxyapatite-Based Composite for Jaw Bone Regeneration
Acronym: Flexi2024
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Pietro Felice, Prof. Pietro Felice, University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG0091421_2024
Record Dates: First submitted 2024-08-07; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Bone Atrophy; Edentulism; Bone Regeneration
Keywords: bone regeneration; dental implants; jaws atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with hydroxyapatite-based composite (Experimental): Patients with partially edentulous and atrophic jaws, requiring implant-prosthetic rehabilitation (from 1 to 3 implants), classified as Seibert Class II or III, and needing a GBR bone regeneration intervention with defects not exceeding 7 mm in height. Patients must be 18 years or older and must provide informed consent.
  Interventions: Device: Placement of resorbable HAp-based composite

INTERVENTIONS:
Device: Placement of resorbable HAp-based composite — The resorbable HAp-based composite device will be immersed in a saline solution for 15 minutes, allowing it to transition from a rigid state to a flexible and deformable one (Fig. 1). Subsequently, the device will be shaped appropriately on the resin model, ensuring proper placement within the bone defect to be regenerated. Patients will receive antibiotic prophylaxis of 1 g amoxicillin, 1 hour before the procedure (or 300 mg clindamycin in case of penicillin allergy). Before the surgical procedure, patients will rinse with 2% chlorhexidine for one minute to reduce the bacterial load in the oral cavity. For the surgical procedure, under local anesthesia with Articaine and Adrenaline 1:100000, mucoperiosteal flaps will be raised. The pre-shaped resorbable device will then be adapted to the defect and fixed with osteosynthesis screws, used according to clinical practice for this type of intervention. Finally, the flaps will be sutured to ensure primary intention closure.

SUMMARY:
Following a review of the scientific literature, it was found that there are no clinical studies but only in vitro and in vivo studies, which show promising results in terms of bone formation and integration. However, it is necessary to evaluate how well the regenerated bone maintains its structural integrity over time, considering masticatory function and real-life biomechanics. Factors such as mechanical load, remodeling dynamics, and interactions with surrounding tissues could influence the long-term stability of the regenerated bone. Additionally, another important aspect to study is the potential complications and adverse effects associated with the use of the flexible HAp-based composite.

DETAILED DESCRIPTION:
Following a review of the scientific literature, it was found that there are no clinical studies but only in vitro and in vivo studies, which show promising results in terms of bone formation and integration. However, it is necessary to evaluate how well the regenerated bone maintains its structural integrity over time, considering masticatory function and biomechanics in real-life scenarios. Factors such as mechanical load, remodeling dynamics, and interactions with surrounding tissues could influence the long-term stability of the regenerated bone. Additionally, another important aspect to study is the potential complications and adverse effects associated with the use of the flexible HAp-based composite.

Study Objectives The primary objective is to evaluate the efficacy in terms of regenerated bone volume using the new flexible HAp-based composite in mixed bone defects of the jawbones.

Primary Outcome Measures The volume of regenerated bone will be measured using CBCT scans before device placement, immediately after the surgical procedure, and at 8 months post-procedure. The percentage of regenerated bone obtained compared to the initially planned augmentation, i.e., the mean volume difference, will be calculated before the surgical procedure, immediately after device placement, and at 8 months.

Secondary Objectives These include evaluating intraoperative and postoperative complications occurring at the time of placement or after device placement, assessing the conditions of peri-implant hard and soft tissues, measuring overall patient satisfaction with the treatment, analyzing the correlation between implant survival and various systemic and clinical patient factors, and conducting a histological evaluation of vascularization and new bone formation in samples of regenerated bone taken during implant site preparation.

Secondary Outcome Measures The condition of hard tissues will be assessed based on periapical intraoral radiographs. For soft tissue conditions, for each implant site, peri-implant probing depth (PPD), bleeding on probing (BOP), presence of peri-implant plaque (mPLI), and the amount of keratinized gingiva will be considered at m3, m6, m9, and m12 from implant placement. Any pathological events such as neurological lesions, exposures, infections, inflammation, fractures, or loosening of prosthetic screws, and prosthesis fractures reported in the clinical record during or after device placement and throughout the clinical follow-up will be evaluated as outcomes of intraoperative and postoperative complications at m3, m6, m9, and m12 from device placement. To evaluate overall patient satisfaction, two validated questionnaires will be analyzed: the Oral Health Impact Profile (OHIP-14) and a Patient Satisfaction questionnaire. To assess the correlation between implant survival and certain systemic and clinical patient factors, the following independent variables will be studied: age, gender, smoking status, jaw in which the implants were placed, type of implant, implant length, implant diameter, and compared with implant survival data. Histological and histomorphometric analysis will be conducted on samples of regenerated bone collected during implant site preparation at the passage of the first preparation drill.

Study Plan A total of 20 patients will be included in the study.

Study Design This is a spontaneous, prospective, interventional clinical investigation with post-marketing medical device analysis, enrolling patients with jaw bone atrophy at the Oral Surgery Unit of the Dental Clinic, University of Bologna. Collaboration with the laboratory at the University of Chieti-Pescara, Department of Medical, Oral, and Biotechnological Sciences, is planned. Insurance will be covered by university funds for Oral Surgery.

Study Start Date/Enrollment: After Ethics Committee approval and obtaining corporate clearance Prospective Period: 1 year Total Study Duration: 5 years (including individual follow-ups and data processing)

Study Population Inclusion Criteria Patients with partially edentulous and atrophic jaws, requiring implant-prosthetic rehabilitation (from 1 to 3 implants), classified as Seibert Class II or III, and needing a GBR bone regeneration intervention with defects not exceeding 7 mm in height. Patients must be 18 years or older and must provide informed consent.

Exclusion Criteria General contraindications to implant surgery. Patients who have received head and neck irradiation of more than 70 Gray. Immunocompromised and immunosuppressed patients. Patients treated or under treatment with intravenous amino-bisphosphonates. Patients with poor oral hygiene and motivation. Uncontrolled diabetes. Pregnancy or breastfeeding. Drug or alcohol dependency. Psychiatric conditions that contraindicate surgical treatment. Limited mouth opening (less than 3.5 cm between the two arches in the anterior region). Patients with acute or chronic inflammation/infection at the implant site. Patients referred solely for implant placement.

Medical Device Under Study The study focuses on a bio-composite bone substitute based on hydroxyapatite (Flexi-Oss, Medical Inventi S.A., Lublin, Poland). This is a biphasic material comprising hydroxyapatite and a polymer component.

Statistical Methods Sample Size The mean regenerated bone volume using a semi-occlusive CAD/CAM titanium device from a previous study was 1524 mm³. Considering an estimate of 1380 mm³ of regenerated bone using the hydroxyapatite-based bio-composite bone substitute, with a standard deviation of 200 mm³, a significance level (alpha) of 0.05, and a statistical power of 80%, using the two-sided Z test, it was determined that 16 patients need to be enrolled. Considering a potential dropout rate of 20%, the number of patients to be included in the study has been increased to 20.

ELIGIBILITY:
Inclusion Criteria:

* Patients with partially edentulous and atrophic jaws, requiring implant-prosthetic rehabilitation (from 1 to 3 implants), classified as Seibert Class II or III, and needing a GBR bone regeneration intervention with defects not exceeding 7 mm in height
* Age 18 years or older
* Obtaining informed consent

Exclusion Criteria:

* Patients who have received radiation therapy to the head and neck with more than 70 Gray.
* Immunocompromised and immunosuppressed patients.
* Patients treated with or currently receiving intravenous amino-bisphosphonates.
* Patients with poor oral hygiene and lack of motivation.
* Uncontrolled diabetes.
* Pregnancy or breastfeeding.
* Drug or alcohol dependence.
* Psychiatric conditions that contraindicate surgical treatment.
* Limited mouth opening (less than 3.5 cm distance between the two arches in the anterior area).
* Patients with acute or chronic inflammation/infection at the implant site.
* Patients referred solely for implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Regenerated Bone Volume | From the treatment and after 8 months,
  he volume of regenerated bone will be measured using CBCT scans before device placement, immediately after the surgical procedure, and at 8 months post-procedure. The percentage of regenerated bone obtained compared to the initially planned augmentation, i.e., the mean volume difference, will be calculated before the surgical procedure, immediately after device placement, and at 8 months. It is specified that CBCT scans and the procedure are performed as part of routine clinical practice.

SECONDARY OUTCOMES:
Complications | Months 1, 3, 6, 8, and 12.
  Any pathological events such as neurological lesions, exposures or infections of the placed medical device, inflammation, fractures or loosening of prosthetic screws, prosthesis fracture, etc., reported in the clinical record and occurring during or after implant placement and throughout the clinical follow-up (m1; m3; m6; m8; and m12 from the surgical placement of the device) will be evaluated as outcomes of intraoperative and postoperative complications.
Patient Satisfaction | At 1 month and 9 months after treatment
  To evaluate the overall satisfaction of patients undergoing the treatment, a validated questionnaire, the Oral Health Impact Profile (OHIP-14), is completed by patients during follow-up visits. The same questionnaire will be administered to patients one month after the surgical procedure and eight months after the procedure. OHIP is a 14-item questionnaire.
Correlation between implant survival and certain systemic and clinical patient factors | After Treatment for 3 years
  The following independent variables will be studied: age, gender, smoking status, jaw in which the implants were placed, type of implant, implant length, implant diameter, and compared with implant survival data (m6, m12, and 3 years)
Histological analysis | 8 months after device placement.
  Histological analysis on samples of regenerated bone collected during the preparation of the implant site, specifically during the passage of the first preparation drill. Paraffin sections will be cut at 4 µm, fixed in formalin, and mounted on slides treated with 3-aminopropyltriethoxysilane. The sections will then undergo immunostaining for blood vessels using antibodies against CD31, VEGF, and KDR epitopes.The criteria established by Weidner and Folkman will be used to identify blood vessels in the immunostained sections. Specifically, positively stained endothelial cells or groups of endothelial cells, regardless of shape and size, that are clearly separated from adjacent blood vessels or other connective tissues, will be counted as blood vessels. Vascular nodules, although usually present, will not be considered a definition of a blood vessel, and red blood cells will not be used to calculate the vascular lumen.
Hard Tissues Conditions | At months: 3, 6, 12 and 3 years after treatment
  The condition of hard tissues is assessed based on periapical intraoral radiographs, taken using the parallel technique before and after the preservation procedure, at the time of implant placement, at the initial loading, and at the final prosthetic loading and various follow-ups.
Peri-implant probing depth (PPD) in mm | At months: 3, 6, 12 and 3 years after treatment
  The condition of soft tissues is evaluated using periodontal indices and recorded in the clinical record: using a periodontal probe, the peri-implant probing depth (PPD) will be evaluated in millimiters, and the are measured for each implant site (at m3, m6, m12, and 3 years post-implant placement).
bleeding on probing (BOP), | At months: 3, 6, 12 and 3 years after treatment
  Using a periodontal probe, the presence of bleeding around the implants will be recorded in the clinical record.
Amount of keratinized gingiva | At months: 3, 6, 12 and 3 years after treatment
  Using a periodontal probe, the amount of keratinized gingiva will be assessed in millimiters and recorded in clinical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinic, Unit of Oral Surgery, University of Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Original articles in international journals
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From September 2025
Access Criteria: Access credentials to journal resources
URL: https://docs.google.com/document/d/10_Zx-mAGhn2yLDdFFHMerulRq43RDyLO7sXjScR6auc/edit?pli=1